CLINICAL TRIAL: NCT04959669
Title: Effectiveness of an Electronic Decision Support System (DeSSBack) in Improving the Management of Low Back Pain: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of an Electronic Decision Support System (DeSSBack) in Improving the Management of Low Back Pain
Acronym: DeSSBack
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Teo Chin Hai, Senior Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PV041-2019
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual care
- Intervention group (Experimental): DeSSBack (Decision Support System for Low Back Pain)
  Interventions: Other: DeSSBack

INTERVENTIONS:
Other: DeSSBack — The DeSSBack (Decision Support System for Low Back Pain) is a decision support tool developed in the University of Malaya Medical Centre's (UMMC) electronic medical record system by adopting and re-packaging the STaRT system to suit the local context. It stratifies patients with low back pain to low, medium or high risk, which are then managed differently. The DeSSBack has also been incorporated the local clinical practice guidelines and feedback from local experts.
  Arms: Intervention group

SUMMARY:
Low back pain is a common health problem where over than half a billion people worldwide suffers from it. In Malaysia, back pain is among the top ten reasons why people see a doctor. Although there are many guidelines available, healthcare professionals still find managing low back pain as challenging.

The Decision Support System for Low Back Pain (DeSSBack) has been developed by adopting and re-packaging STaRT system, incorporate with the local clinical practice guidelines and feedback from local experts. It aims to aid healthcare professionals in managing low back pain through a stratified approach.

The objective of the study is to evaluate the effectiveness of DeSSBack in improving the management of patients with low back pain in a primary care clinic. We hypothesise that the implementation of DeSSBack will improve the outcomes of low back pain patients including quality of life, emotional state and level of pain.

This study protocol presents the rationale and design of a cluster randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking care for low back pain at the primary care clinic in UMMC
* Male and female
* Age 18 years and above
* Can understand Malay and English

Exclusion Criteria:

* Potentially serious pathology (eg: cauda equina compression, inflammatory arthritis, malignancy and etc)
* Serious co morbidity
* Psychiatric illness or personality disorder
* Spinal surgery in the last 6 months
* Pregnant
* Already receiving treatment other than primary care for this episode of back pain
* Inability to attend regular physiotherapy appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in health status measure for low back pain between baseline and 2-month | Baseline, 2-months
  We are measuring the changes in health status with Rolland Morris Disability Questionnaire (RMDQ). The score ranges from a minimum of 0 to a maximum of 24. Greater levels of disability are reflected by higher scores.
Changes in health status measure for low back pain between baseline and 6-month | Baseline, 6-months
  We are measuring the changes in health status with Rolland Morris Disability Questionnaire (RMDQ). The score ranges from a minimum of 0 to a maximum of 24. Greater levels of disability are reflected by higher scores.

SECONDARY OUTCOMES:
Changes in the Hospital Anxiety and Depression Scale (HADS) between baseline and 2-month | Baseline, 2-months
  The HADS is a self-assessment questionnaire to assess states of anxiety and depression in the setting of hospital outpatient clinic. The minimum value is 0 and the maximum value is 21 for both anxiety and depression. The higher the score, the worse the outcome is.
Changes in the Hospital Anxiety and Depression Scale (HADS) between baseline and 6-month | Baseline, 6-months
  The HADS is a self-assessment questionnaire to assess states of anxiety and depression in the setting of hospital outpatient clinic. The minimum value is 0 and the maximum value is 21 for both anxiety and depression. The higher the score, the worse the outcome is.
Changes in the back pain severity score between baseline and 2-month | Baseline, 2-months
  The back pain severity score is a self-assessment score to rate severity of the back pain. Patients would rate their back pain from 0 being no pain at all, to 10 being unbearable pain.
Changes in the back pain severity score between baseline and 6-month | Baseline, 6-months
  The back pain severity score is a self-assessment score to rate severity of the back pain. Patients would rate their back pain from 0 being no pain at all, to 10 being unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Tun Firzara AM, Teo CH, Teh SY, Su JY, Mohd Zaini HS, Suhaimi A, Ng WL, Danaee M, Stevenson K, Mallen CD, Ng CJ. Evaluation of an electronic clinical decision support system (DeSSBack) to improve low back pain management: a pilot cluster randomized controlled trial. Fam Pract. 2023 Dec 22;40(5-6):742-752. doi: 10.1093/fampra/cmad044. PMID 37237425